CLINICAL TRIAL: NCT03228069
Title: Humoral and Cell-mediated Immune Responses and Immunological Tolerance After Rabies Booster Vaccination in Previously Rabies Immunized HIV-infected Adults
Brief Title: Immune Responses and Immunological Tolerance After Rabies Booster Vaccination in HIV-infected Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen Saovabha Memorial Institute (Other)
Responsible Party: Principal Investigator, Suda Sibunruang, Medical doctor, Queen Saovabha Memorial Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1/2017
Record Dates: First submitted 2017-07-14; First posted 2017-07-24 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Rabies
Keywords: rabies vaccination
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Intervention Model Description: The volunteers who participated in the previous clinical trials were invited to join this study. Of which, there were 2 groups, one received a single visit 4-site intradermal rabies booster vaccination. The another received a conventional intramuscular rabies booster vaccination on day 0 and 3.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single visit 4-site ID vaccination (Experimental): Blood would be drawn from those who received a single visit 4-site ID rabies booster vaccination in the previous trial.
  Interventions: Procedure: Blood drawn after rabies booster vaccination
- Conventional IM vaccination (Active Comparator): Blood would be drawn from those who received a conventional intramuscular rabies booster vaccination in the previous trial.
  Interventions: Procedure: Blood drawn after rabies booster vaccination

INTERVENTIONS:
Procedure: Blood drawn after rabies booster vaccination — Blood would be drawn for testing of rabies neutralizing antibody titers, rabies specific T lymphocytes and regulatory T cells after receipt of rabies booster vaccination at least a year before.

SUMMARY:
To study the humoral and cell-mediated immune responses in HIV-infected adults who had previously received rabies booster vaccination more than a year before

DETAILED DESCRIPTION:
Previous study has shown the higher immunogenicity response among HIV-infected adults who received a single visit 4-site intradermal rabies booster vaccination than those who received the conventional intramuscular regimen. The investigators follow the persistence of these effects. Also, the regulatory T cell levels were examined after the rabies booster vaccination .

ELIGIBILITY:
Inclusion Criteria:

* Healthy HIV-infected adults
* Previously received rabies booster vaccination by participation in the previous clinical trials of the investigators.

Exclusion Criteria:

* Have any active opportunistic infections
* Received blood or blood product within 3 months
* Received anti-malarial drugs
* Received rabies vaccination in a previous year.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Rabies Neutralizing Antibody Titers (RNab) | GMTs of RNab and proportion of volunteers who have had RNab above protective antibody levels (0.5 IU/ml) after receipt of rabies booster vaccination at least a year before were compared between 2 arms at one time point on the date of study recruitment.
  Rabies Neutralizing Antibody Titers would be represented and compared by geometric mean titers (GMTs)

SECONDARY OUTCOMES:
Rabies specific T cell response | Numbers of spots, of which represent the rabies specific T cell response after receipt of rabies booster vaccination at least a year before were compared between 2 arms at one time point on the date of study recruitment.
  Rabies specific T cell response is measured by Enzyme - linked Immunospot Assay (ELISPOT)

OTHER OUTCOMES:
Rabies specific regulatory T cells | Numbers of Rabies specific regulatory T cells after receipt of rabies booster vaccination at least a year before were compared between 2 arms at one time point on the date of study recruitment.
  Rabies specific regulatory T cells is measured by flow cytometry method

CONTACTS AND LOCATIONS:
Overall Officials: Suda Sibunruang, MD, Principal Investigator — Queen Saovabha Memorial Institute
Locations (1):
- Queen Saovabha Memorial Institute, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No